CLINICAL TRIAL: NCT03786146
Title: Changes in Retinal Nerve Fiber Layer Thickness Detected by Optical Coherence Tomography in Diabetic Retinopathy After Panretinal Photocoagulation
Brief Title: Changes in Retinal Nerve Fiber Layer Thickness Detected by OCT in Diabetic Retinopathy After Panretinal Photocoagulation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rania M. Goda, principle investigator, Assiut University
Other Study IDs: RNFL in diabetic after PRP
Record Dates: First submitted 2018-12-14; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Panretinal photocoagulation reduces the risk of visual loss by 50% in patients with diabetic retinopathy. It is recognized that laser expansion into the retina may be associated with photoreceptor loss, retinal pigment epithelial hypertrophy and visual field loss.

Panretinal photocoagulation can cause alteration in retinal vascular permeability therefore, retinal thickness may be increased including retinal nerve fiber layer. On the contrary, it can damage retinal cells including ganglion cells, which may decrease the retinal nerve fiber layer thickness in the latter follow up period.

Peripapillary retinal nerve fiber layer can be measured by optical coherence tomography which is a non-invasive technique for obtaining high resolution cross sectional images of a tissue.

DETAILED DESCRIPTION:
Pre laser assessment:

* Assessment of medical and family history
* Refraction and best corrected visual acuity
* Anterior segment examination using binocular slit lamp bi-microscopy.
* Posterior segment examination.
* OCT scan of peripapillary area

Post laser assessment ( at 1,3 and 6 months):

* Refraction and best corrected visual acuity.
* Anterior segment examination using binocular slit lamp bi-microscopy.
* Posterior segment examination.
* OCT scan of peripapillary area.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of proliferative diabetic retinopathy.
* Treated by panretinal photocoagulation.
* Age between 40-70 years old.

Exclusion Criteria:

* Patients with densely opaque media (as dense cataract or vitreous hemorrhage).
* Glaucomatous patients.
* Any other associated retinopathy.

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be carried out on patients with a clinical diagnosis of proliferative diabetic retinopathy treated by panretinal photocoagulation.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Retinal nerve fiber layer thickness measured by Optical Coherence Tomography (OCT) and expressed in micrometers. | 0 (before laser treatment ).
  A 3.4 mm OCT circular scan will be positioned around the optic nerve head.
Retinal nerve fiber layer thickness measured by Optical Coherence Tomography (OCT) and expressed in micrometers. | 1 month post laser treatment.
  A 3.4 mm OCT circular scan will be positioned around the optic nerve head.
Retinal nerve fiber layer thickness measured by Optical Coherence Tomography (OCT) and expressed in micrometers. | 3 months post laser treatment.
  A 3.4 mm OCT circular scan will be positioned around the optic nerve head.
Retinal nerve fiber layer thickness measured by Optical Coherence Tomography (OCT) and expressed in micrometers. | 6 months post laser treatment.
  A 3.4 mm OCT circular scan will be positioned around the optic nerve head.

CONTACTS AND LOCATIONS:
Overall Officials: rania goda, Principal Investigator — researcher in Assiut university; ehab wasfi, Study Director — Assiut University; Ali Netag, Study Director — Assiut University; Kamel Abd Elnaser, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wagdy F, El Sobky H, Sarhan AE-R, Hafez M. Evaluation of retinal nerve fiber layer thickness in diabetic retinopathy by optical coherence tomography after full scatter panretinal argon laser photocoagulation. J Egypt Ophthalmol Soc [Internet]. 2013 Jul 1;106(3):153-8. Available from: http://www.jeos.eg.net/article.asp?issn=2090-0686
- [Background] Kim HY, Cho HK. Peripapillary retinal nerve fiber layer thickness change after panretinal photocoagulation in patients with diabetic retinopathy. Korean J Ophthalmol. 2009 Mar;23(1):23-6. doi: 10.3341/kjo.2009.23.1.23. Epub 2009 Mar 9. PMID 19337475
- [Background] Kim J, Woo SJ, Ahn J, Park KH, Chung H, Park KH. Long-term temporal changes of peripapillary retinal nerve fiber layer thickness before and after panretinal photocoagulation in severe diabetic retinopathy. Retina. 2012 Nov-Dec;32(10):2052-60. doi: 10.1097/IAE.0b013e3182562000. PMID 23099450
- [Background] Paunescu LA, Schuman JS, Price LL, Stark PC, Beaton S, Ishikawa H, Wollstein G, Fujimoto JG. Reproducibility of nerve fiber thickness, macular thickness, and optic nerve head measurements using StratusOCT. Invest Ophthalmol Vis Sci. 2004 Jun;45(6):1716-24. doi: 10.1167/iovs.03-0514. PMID 15161831
- [Background] Lim MC, Tanimoto SA, Furlani BA, Lum B, Pinto LM, Eliason D, Prata TS, Brandt JD, Morse LS, Park SS, Melo LA Jr. Effect of diabetic retinopathy and panretinal photocoagulation on retinal nerve fiber layer and optic nerve appearance. Arch Ophthalmol. 2009 Jul;127(7):857-62. doi: 10.1001/archophthalmol.2009.135. PMID 19597104
- [Background] Muqit MM, Wakely L, Stanga PE, Henson DB, Ghanchi FD. Effects of conventional argon panretinal laser photocoagulation on retinal nerve fibre layer and driving visual fields in diabetic retinopathy. Eye (Lond). 2010 Jul;24(7):1136-42. doi: 10.1038/eye.2009.308. Epub 2009 Dec 18. PMID 20019760